CLINICAL TRIAL: NCT03475940
Title: Coagulopathy in Cardiac Surgery; a Quaternary-care Academic Center Experience
Brief Title: Coagulopathy in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chaowanan Khamtuikrua, lecturer, Mahidol University
Other Study IDs: Si2018-2
Record Dates: First submitted 2017-12-31; First posted 2018-03-23 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Coagulopathy, Cardiac Surgery, Cardiopulmonary Bypass
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coagulopathy in cardiac surgery; a quaternary-care academic center experience

Objectives:

Primary:

To determine incidence of coagulopathy after cardiac surgery in Thai people To determine incidence of resternotomy for stop bleeding, morbidity and mortality

Secondary:

To identify risk factors which associated with non-red cell transfusion and coagulopathy

study decide: Retrospective chart review

DETAILED DESCRIPTION:
Data to be collected:

Age*, gender* Body weight, height, body mass index* Underlying disease: DM, renal disease*, liver disease* Pre-op. Antiplatelet or anticoagulant* Pre-op coagulogram and platelet count* Emergency or elective surgery Resternotomy or not* Intraoperative blood component Intraoperative factor concentration Dose and timing of antifibrinolytic administration* CPB time* Postoperative body temperature*

*Possible risk factors for non-red cell transfusion

statistic: To assess the relationship between risk factors and non-red cell transfusion a univariate analysis was performed using an unpaired t-test and a Chi-square test.

For higher accuracy regarding the impact of single risk factors, a multiple logistic regression analysis was also performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Schedule to cardiac surgery under cardiopulmonary bypass

Exclusion Criteria:

* Schedule for aortic surgery or complex congenital cardiac surgery
* Using ECMO before surgery
* Incomplete anesthetic record

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 years Schedule to cardiac surgery under cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
incidence of coagulopathy after cardiac surgery in Thai people | 1 year
  coagulopathy and throbocytopenia

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of medicine Siriraj hospital, Bangkok Noi, Bangkok
  - faculty of medicine Siriraj hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No